CLINICAL TRIAL: NCT00532688
Title: Randomised Control Pilot Trial of n-Acetylcysteine in the Treatment of Chronic Heart Failure With Coexistent Chronic Renal Failure.
Brief Title: N-Acetylcysteine in Heart Failure With Coexistent Chronic Renal Failure
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: The Alfred (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 132/07
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Heart Failure, Congestive; Kidney Failure, Chronic
Keywords: acetylcysteine; N-acetylcysteine; heart failure; renal failure
MeSH Terms: conditions — Heart Failure; Kidney Failure, Chronic; Renal Insufficiency | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 5 patients: 28 days of n-acetylcysteine (in addition to standard therapy) and then repeat serum creatinine and vascular study then crossover to placebo for 28 days after one week washout period.
  Interventions: Drug: N-acetylcysteine
- 2 (Placebo Comparator): 28 days of oral distilled water (5ml) (in addition to standard therapy) and then repeat serum creatinine and vascular study then crossover to intervention (N-acetylcysteine 500mg oral bd) for 28 days after one week washout period with tests repeated again at 4 weeks and 9 weeks.
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — 28 days of oral n-acetylcysteine (500mg bd)(in addition to standard therapy) and then repeat serum creatinine and vascular study then crossover to placebo for 28 days after one week washout period with tests repeated again at 4 weeks and 9 weeks.
  Other Names: Mucomyst(R)

SUMMARY:
Treatment with n-acetylcysteine in patients with heart failure and chronic renal failure leads to improvements in vascular function and in renal function.

DETAILED DESCRIPTION:
Ten patients will be invited to participate in the trial. After obtaining informed consent, the ten patients will be randomly assigned to one month of treatment with oral n-acetylcysteine 500mg or placebo twice daily for thirty days in addition to their regular therapy. At enrolment the patients will be educated and counselled about the trial and the intervention medication. Patients will also have a blood test (serum creatinine) that will allow the calculation of their renal function by use of the Cockroft Gault equation. Blood samples will also be frozen and stored. Patients will also undergo an ultrasound test of the function of their arm blood vessels. Both the blood test and the ultrasound test will be repeated at the completion of the thirty day trial period. Again the blood test sample will be frozen and stored. Subjects will then cross over to the other treatment arm for a further one month period, with the same testing at the end.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years inclusive;
* Patients with chronic heart failure NYHA II, III and IV and LVEF<40%. Stable medications for 1 month. Not admitted to hospital in the past month.
* Chronic renal failure with GFR (as estimated by the Cockroft Gault equation) of >30 ml/min and <50 ml/min not on any form of dialysis.

Exclusion Criteria:

* Age <18 and >75 years;
* Myocardial infarction in the preceding six months;
* Acute decompensation of renal function or heart failure in the last 30 days;
* Allergy to n-acetylcysteine or glyceryl trinitrate;
* Contraindications to the use of glyceryl trinitrate as per the product information lodged with the PBS (Australia);
* On treatment with allopurinol, vitamin C or vitamin E or other antioxidant therapy at time of randomisation (statins are acceptable);
* Acute decompensation of another organ system in the last 30 days;
* Current pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-09; Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
Vascular function via non invasive ultrasound measured flow mediated dilatation | baseline, 4 weeks and 9 weeks
Estimated glomerular filtration rate calculated with Cockroft Gault equation. | baseline, 4 weeks, 9 weeks

SECONDARY OUTCOMES:
Symptoms of heart failure | baseline, 4 weeks, 9 weeks
Death | baseline, 4 weeks, 9 weeks
Serum BNP (brain natriuretic peptide) | baseline, 4 weeks, 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Kaye, PhD FRACP, Principal Investigator — Alfred Heart Centre; Anthony Camuglia, MBBS, Principal Investigator — The Alfred; Catherine Farrrington, Principal Investigator — Alfred Heart Centre; Jenny Starr, Principal Investigator — Alfred Heart Centre
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Camuglia AC, Maeder MT, Starr J, Farrington C, Kaye DM. Impact of N-acetylcysteine on endothelial function, B-type natriuretic peptide and renal function in patients with the cardiorenal syndrome: a pilot cross over randomised controlled trial. Heart Lung Circ. 2013 Apr;22(4):256-9. doi: 10.1016/j.hlc.2012.10.012. Epub 2012 Dec 7. PMID 23219310